CLINICAL TRIAL: NCT04194684
Title: Nab-Paclitaxel in Patients With ER+/HER2- Recurrent Metastatic Breast Cancer：a Multi-center Study
Brief Title: Nab-Paclitaxel in Patients With ER+/HER2- Recurrent Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2129
Record Dates: First submitted 2019-12-10; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): Nab-paclitaxel
  Interventions: Drug: nab-paclitaxel

INTERVENTIONS:
Drug: nab-paclitaxel — nab-paclitaxel 125mg / m2, intravenous drip 30min, d1, 8, 21 days as a cycle, until the disease progresses or intolerable toxicity. According to the calculation results, the administered dose can be within ± 10% of the calculated dose.

SUMMARY:
This study is a single-arm, open, multi-center clinical study of nab-paclitaxel as the therapy ER+/HER2- recurrent metastatic breast cancer。

ELIGIBILITY:
Inclusion Criteria:

1. Female, 18 to 70 years old;
2. histologically confirmed recurrent or metastatic breast cancer, ER-positive (> 10%), HER-2 negative (Definition: immunohistochemical [IHC] 0, 1+, or in situ hybridization [ISH] negative It is defined as the ratio of HER2 gene copy number to the number of CEP17 signals is less than 2.0, or for single probe detection, the HER2 gene copy number is less than 6);
3. After transfer, ≤2 lines and ≥1 line endocrine therapy, and progress;
4. at least one measurable lesion according to RECIST 1.1 ;
5. ECOG score≤2;
6. Expected survival≥3 months;
7. Bone marrow function: white blood cells≥3×109/L, neutrophils≥1.5×109/L, platelets ≥100×109 / L, hemoglobin≥90g / L;
8. Liver and kidney function: total bilirubin (TBIL) ≤1.5 times the upper limit of normal value, alanine aminotransferase (ALT), aspartate aminotransferase (AST) are ≤2.5 times the upper limit of normal value; if due to liver metastasis, the above indicators ≤5 times the upper limit of normal value; serum creatinine (Cr) ≤1.5 times the upper limit of normal value;
9. taxane adjuvant chemotherapy for more than 1 year;
10. Women of childbearing age have a negative pregnancy test and must agree to take effective contraceptive measures during the study and within 3 months after the last dose
11. Sign written informed consent before the test.

Exclusion Criteria:

1. Received chemotherapy after transfer;
2. Patients with congestive heart failure with a grade II or above identified by the New York Heart Association (NYHA) score;
3. Uncontrolled brain metastases;
4. Severe systemic infections;
5. Peripheral neuropathy of degree II or above within 4 weeks before enrollment, or patients known to be allergic or intolerant to this drug;
6. Important organ diseases:liver and kidney dysfunction, history of myocardial infarction, unstable heart disease, chronic active hepatitis, etc .;
7. History of other malignant tumors within 5 years (except cured cervical cancer or skin basal cell carcinoma);
8. Received other anti-tumor treatments or other experimental drugs within 1 month before starting treatment;
9. Patients participating in other clinical trials at the same time;
10. Any medical condition in which the investigator considers the patient unsuitable for study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-12-28 (Estimated); Primary Completion 2022-12-28 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Estimated up to 1 year
  Defined as proportion of complete response and partial response according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Clinical benefit rate | CR+PR+SD≥8 weeks
  Defined as proportion of complete response 、partial response and stable disease according to RECIST 1.1 criteria.
Progression-Free Survival (PFS) | Estimated up to 2 year
  Calculated from the time the study drug was first administered to the first confirmation of disease progression or death (whichever occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No